CLINICAL TRIAL: NCT02371928
Title: A Neuromuscular Exercise Program for Patients With Anterior Shoulder Instability: A Randomized Controlled Trial
Brief Title: A Neuromuscular Exercise Program for Patients With Anterior Shoulder Instability
Acronym: SINEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); The Danish Rheumatism Association (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Eshoj, Msc, PhD. stud, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20140093
Record Dates: First submitted 2015-02-09; First posted 2015-02-26 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Shoulder Dislocation; Musculoskeletal Diseases
Keywords: Shoulder; Instability; Neuromuscular; Physiotherapy; Exercise; Dislocation; Recurrence
MeSH Terms: conditions — Shoulder Dislocation; Musculoskeletal Diseases; Motor Activity; Joint Dislocations; Recurrence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular exercise program (Active Comparator): A 12-week physiotherapeutic, supervised exercise program with focus on neuromuscular shoulder control besides incorporation of kinetic chain exercises.
  The exercise program contains the following focal points: Scapula and glenohumeral setting/control, dynamic shoulder stability, muscle co-contractions (weight-bearing upper extremity exercises) and proprioceptive training.
  Interventions: Other: Neuromuscular exercise program
- Standard home exercise program (Active Comparator): One physiotherapeutic-supervised instruction in 12 weeks of active exercises for the rotator cuff and scapular muscles.
  Information about the shoulder injury and how to avoid pain provoking movements besides future implications is given. Also, participants receives one phone call after six weeks of training from a physiotherapist to ensure good compliance and answer any questions that the patient may have.
  Interventions: Other: Standard home exercise program

INTERVENTIONS:
Other: Neuromuscular exercise program — Exercises can be individually progressed from basic to elite level.
  Low load exercises are performed every day with 2 sets of 20-25 repetitions whereas high load exercises are performed three times per week with 2 sets of 8-12 repetitions.
  Exercises are progressed using the following components: arm-position, load, speed, open/closed eyes, stable/unstable surfaces.
  Patients have online access to instructions and video recordings of all exercises and progression levels. Patients are trained to continuously evaluate their own shoulder function and to adjust the exercise levels themselves at home.
  Supervision will be given two times a week for the first two weeks and then once a week for the remaining period.
  Arms: Neuromuscular exercise program
Other: Standard home exercise program — Strengthening of the rotator cuff muscles are performed with the use of elastic bands (shoulder internal and external rotation besides abduction in scapular plane) whereas mobility/strengthening exercise for the scapular muscles are performed through weight-bearing positions and movements of the upper extremity.
  All exercises are performed three times a week with 2 sets of 10 repetitions.
  Arms: Standard home exercise program

SUMMARY:
This study is designed to investigate the efficacy and safety of a supervised neuromuscular exercise program versus a standard home exercise program for patients with post-traumatic symptomatic anterior shoulder instability.

Participants with at least one week of symptom duration are randomly assigned to either a 12-week structured, supervised Shoulder Instability Neuromuscular EXercise (SINEX) program versus a standard HOMe EXercise (HOMEX) program.

The H1-hypothesis is that the SINEX program results in a greater increase in quality of life and physical function than the HOMEX program at the primary endpoint at three months follow-up from baseline

DETAILED DESCRIPTION:
A common, and very painful, injury for individuals in their second and third decades is a traumatic dislocated shoulder. This injury accounts for almost 50% of all joint dislocations registered in the emergency departments. Due to post-traumatic laxity and injuries to the surrounding shoulder tissue, one major problem is the risk of developing a chronic recurrent instable shoulder affecting patients both physically and psychologically decreasing their overall quality of life.

Biomechanically, proprioceptive changes and decreased sensorimotor control are found in patients with post-traumatic shoulder instability inhibiting the ability to control and stabilize the glenohumeral joint. In other similar musculoskeletal disorders, recent studies clearly shows positive effects of progressive neuromuscular exercise.

Finally, no studies have yet investigated the effect of a structured, physical exercise-training regime based on neuromuscular principles targeting the shoulder joint.

This trial is performed as a randomized, assessor-blinded, controlled multi-center trial with cooperation from various shoulder outpatient clinics located at different hospitals in The Region of Southern and Northern Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-39
2. Minimum one radiographic verified anterior shoulder dislocation (total dissociation of the humeral head to the glenoid)
3. Limited ability to maintain a desired level of physical activity (sports/leisure/work) due to pain and/or symptoms in the affected shoulder within the latest week.

Exclusion Criteria:

1. Humeral fracture and/or bony bankart (visible on conventional radiographs at the time of presentation) warranted for surgery decided by the orthopedic (no other axial or appendicular musculoskeletal injury)
2. Prior surgery in affected shoulder joint
3. >5 anterior shoulder dislocations (verified by journal or subjective evaluation)
4. Suspected competing diagnosis (e.g. rheumatoid arthritis, cancer, neurological disorders, fibromyalgia, schizophrenia, suicidal threatened, borderline personality disorder or obsessive compulsive disorder
5. Sensory and motor deficits in neck and shoulder
6. Pregnancy
7. Inadequacy in written and spoken Danish
8. Not willing or able to attend 12 weeks of supervised exercise therapy

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Shoulder Instability Index (WOSI) | Primary: 3 months. Other: 12, 24 months
  The patient reported outcome, WOSI, consists of four domains covering "Physical Symptoms", "Sport/Recreation/Work", "Lifestyle" and "Emotions" with 21-item questionnaires in all. Each item is scored using a horizontal visual scale ranging from 0 to 100 mm (0-2100, with 0 as the level of no trouble).

SECONDARY OUTCOMES:
Change in Euro Qol 5D Index (EQ-5D) | 3,12, 24 months
  Quality of life questionnaire
Change in Tampa Scale of Kinesiophobia | 3,12, 24 months
  Fear of movement and re-injury questionnaire
Change in the four sub-scales (domains) of WOSI | 3,12, 24 months
  Questionnaire
Change in Patient Specific Functioning Scale | 3 months
  Questionnaire
Global Perceived Effect | 3 months
  Questionnaire
Change in Constant-Murley Shoulder Score | 3 months
  100-point scoring system with self-reported and objective measurements included.
Number of changes in positive clinical tests for anterior shoulder instability | 3 months
  Provocative clinical tests for anterior shoulder instability will be used to measure the number of positive and negative tests (Apprehension, relocation, surprise test)
Change in shoulder joint position sense | 3 months
  Re-positioning test of the affected shoulder in abduction and flexion with the use of laser pointer measurements.
Number of participants with adverse events | 3 months
  Open-probe questioning at 3 months follow-up besides any adverse events during the 12-week exercise program registered by the physiotherapists supervising the patients.

OTHER OUTCOMES:
Baseline demographics and other relevant information (age, sex, symptom intensity and duration, number of shoulder dislocations, medical use, prior physical treatment, Time to return to sport or work, ) | Baseline and 3,12, 24 months
  Questionnaire
Change in mechanical allodynia (exploratory) | 3 months
  Pain pressure threshold measured in the affected shoulder using a handheld algometer (Algometer Type II) at four sites (m. pec. major, the deltoid m., m. trapezius superior and m. levator scapula) and one site at opposite m. tibialis anterior.
Change in number of sites with pain (exploratory) | 3 months
  Self-reported pain registration within the previous 24 hours shaded on a region-divided body chart.
Change in pain scores | 3, 12, 24 months
  Using 100 mm visual analogue scale (VAS) with anchor points "no pain" and "worst imaginable pain" in various situations.
Change in maximum isometric muscle strength | 3 months
  Measured bilaterally in 90 degrees of abduction in the scapular plane using an Isoforce dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Eshoj, PhD-student, Principal Investigator — Research Unit for Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark; Birgit Juul-Kristensen, Ass. Prof, Study Chair — Research Unit for Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark; Karen Søgaard, Prof., Study Chair — Research Unit for Physical Activity and Health in Working Life, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark; Lars H Frich, MD, Study Chair — Shoulder sector, Orthopaedic Department, Odense University Hospital, Denmark; Steen L Jensen, MD, Study Chair — Shoulder sector, Orthopedic Department, Aalborg University Hospital, Farsø Hospital, Denmark; Sten Rasmussen, MD, Study Chair — Department of Clinical Medicine, Aalborg University, Aalborg, Denmark
Locations (4):
- Denmark (4):
  - Odense University Hospital, Odense, Fyn
  - Aalborg University Hospital, Aalborg, Jutland
  - Hospital of Southwest Denmark, Esbjerg, Jutland
  - Himmerland Hospital, Farsø, Jutland

REFERENCES:
- [Background] Gibson K, Growse A, Korda L, Wray E, MacDermid JC. The effectiveness of rehabilitation for nonoperative management of shoulder instability: a systematic review. J Hand Ther. 2004 Apr-Jun;17(2):229-42. doi: 10.1197/j.jht.2004.02.010. PMID 15162108
- [Background] Handoll HH, Hanchard NC, Goodchild L, Feary J. Conservative management following closed reduction of traumatic anterior dislocation of the shoulder. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004962. doi: 10.1002/14651858.CD004962.pub2. PMID 16437506
- [Background] Zech A, Hubscher M, Vogt L, Banzer W, Hansel F, Pfeifer K. Neuromuscular training for rehabilitation of sports injuries: a systematic review. Med Sci Sports Exerc. 2009 Oct;41(10):1831-41. doi: 10.1249/MSS.0b013e3181a3cf0d. PMID 19727032
- [Background] Robinson CM, Seah M, Akhtar MA. The epidemiology, risk of recurrence, and functional outcome after an acute traumatic posterior dislocation of the shoulder. J Bone Joint Surg Am. 2011 Sep 7;93(17):1605-13. doi: 10.2106/JBJS.J.00973. PMID 21915575
- [Derived] Eshoj HR, Rasmussen S, Frich LH, Hvass I, Christensen R, Boyle E, Jensen SL, Sondergaard J, Sogaard K, Juul-Kristensen B. Neuromuscular Exercises Improve Shoulder Function More Than Standard Care Exercises in Patients With a Traumatic Anterior Shoulder Dislocation: A Randomized Controlled Trial. Orthop J Sports Med. 2020 Jan 30;8(1):2325967119896102. doi: 10.1177/2325967119896102. eCollection 2020 Jan. PMID 32064291
- [Derived] Eshoj H, Rasmussen S, Frich LH, Hvass I, Christensen R, Jensen SL, Sondergaard J, Sogaard K, Juul-Kristensen B. A neuromuscular exercise programme versus standard care for patients with traumatic anterior shoulder instability: study protocol for a randomised controlled trial (the SINEX study). Trials. 2017 Feb 28;18(1):90. doi: 10.1186/s13063-017-1830-x. PMID 28245853